CLINICAL TRIAL: NCT05463211
Title: Quantifying the User Experience, as Well as Neural, Muscular, and Functional Gait Changes Following Exoskeleton-powered Gait Rehabilitation in Children With Mobility Impairments
Brief Title: Exoskeleton-assisted Physiotherapy for Children With Mobility Impairments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: REB 0523
Record Dates: First submitted 2022-06-08; First posted 2022-07-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy
Keywords: Pediatric exoskeleton; Robot assisted gait therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trexo Plus Pediatric Exoskeleton (Experimental): Experimental lower-limb wearable pediatric exoskeleton used biweekly in clinical and school settings.
  Interventions: Device: Trexo Plus Pediatric Exoskeleton

INTERVENTIONS:
Device: Trexo Plus Pediatric Exoskeleton — Wearable pediatric robotic walker for the lower extremities

SUMMARY:
Non-ambulatory children with cerebral palsy (CP) and similar childhood-onset neuromotor conditions face many challenges to fulsome participation in everyday life. Recent initial phase research suggests that physiotherapy paired with use of robotic exoskeletons, such as the Trexo exoskeleton ("The Trexo"; Trexo Robotics, Canada) provides a novel opportunity for children with severe mobility challenges to experience active walking that is individualized to their movement potential (guiding and powering leg movements) and upright support needs. This before-and-after study will assess the first-time experience of 10 non-ambulatory children (ages 4-7) using the Trexo for 6 weeks of twice weekly physiotherapy sessions, and evaluate associated brain, muscle and functional outcomes including accomplishment of individualized goals. To study clinical utility, we will simultaneously capture physiotherapists' (PTs) and PT assistants' (PTAs) training/learning/user experiences with the Trexo's first time use within our center's out-patient program and on-site affiliated school.

This project will contribute evidence-based knowledge to guide clinical decisions about introduction of the Trexo within pediatric rehabilitation settings (target demographic, potential goals, integration into physiotherapy) and be a foundation for a progressive program of multi-centre research. Overall, we hope that this research will lead to better opportunities for children's meaningful participation within the community, including family and peers.

ELIGIBILITY:
Inclusion Criteria:

* Weight of 50-100 lbs (23- 46 kgs), leg length (hip to floor): 40-56c
* GMFCS Level IV equivalent
* Knee and hip range of motion sufficient to allow exoskeleton fit (see exclusion criteria)
* Able to follow GMFM testing instructions, and able to participate in a minimum of 30 minutes of active PT
* Able to reliably signal pain, fear and discomfort
* At least 2 months after any lower limb Botulinum Toxin (BTX) injections
* Will be safe for BTX to be put on hold during their study participation (i.e., a period of 6 months which is equivalent to one BTX treatment cycle).

Exclusion Criteria:

* Any weightbearing restrictions
* Fixed knee contracture (passive) > 20 degrees, knee valgus >40 degrees such that orthosis will not be adaptable to lower limbs. Note: Fixed hip and ankle contractures in themselves are not a contraindication for Trexo
* Hip subluxation > 40% unless with orthopedic clearance for weight bearing with the Trexo
* Orthopaedic surgery within the last 9 months (if muscle) or 12 months (if bone)
* Severe spasticity may be a contraindication (still OK to consider)
* Seizure disorder that is not controlled by medication. For a child on seizure medication, must not have had a seizure in the last 12 months (as verified by the child's treating physician)
* Open skin lesions or vascular disorder of lower extremities
* Osteogenesis imperfecta
* Not able to co-operate for positioning/adjustments within the Trexo
* Involved in another intervention study (any type). May be concurrently enrolled though in a single point assessment study (e.g., annual follow-up of status, measurement study)

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM)-88 - changes from Baseline | Baselines, following 6 weeks of intervention, 1 month post-intervention
  Standard for measuring gross motor skills in children with CP and related neuromotor disorders
Mechanomyography (MMG) - changes from Baseline | Baselines, following 6 weeks of intervention, 1 month post-intervention
  Non-invasive acoustic skeletal muscle recordings (frequency and amplitude)
Structural Magnetic resonance Imaging (MRI) - changes from Baseline | Baseline, following 6 weeks of intervention, 1 month post-intervention
  T1 anatomical scan - grey and white matter volumes
Diffusion Magnetic resonance imaging (MRI) - changes from Baseline | Baseline, following 6 weeks of intervention, 1 month post-intervention
  Multi shell diffusion imaging - kurtosis fractional anisotropy measures
Resting State Functional Magnetic resonance imaging (MRI) - changes from Baseline | Baseline, following 6 weeks of intervention, 1 month post-intervention
  Whole-brain analysis based on BOLD signal changes
Canadian Occupational Performance Measure (COPM) - changes from Baseline | Weekly check-ins for 6 weeks
  Parent reported qualitative questionnaire for gait related goals
Goal Attainment Scaling (GAS) - changes from Baseline | Weekly check-ins for 6 weeks
  Physiotherapist reported qualitative questionnaire for gait related goals; scored -2 to +2

SECONDARY OUTCOMES:
Passive range of motion (ROM) - changes from Baseline | Baselines, following 6 weeks of intervention, 1 month post-intervention
  Range of motion with selected movements measured by the Tardieu Spasticity Scale
Directional Mobility Assessment (DMA) - changes from Baseline | Baselines, following 6 weeks of intervention, 1 month post-intervention
  Simple 10-item functional walking course; scoring key from 0-4
The Sitting Assessment for Children with Neuromotor Dysfunction (SACND) - changes from Baseline | Baselines, following 6 weeks of intervention, 1 month post-intervention
  Evaluates postural tone, proximal stability, postural alignment and balance in sitting on a scale of 1-4
PEDI-CAT Questionnaire - changes from Baseline | Baselines, following 6 weeks of intervention, 1 month post-intervention
  Qualitative parent-report for child's physical and social communication function domains

CONTACTS AND LOCATIONS:
Overall Officials: Tom Chau, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Virginia Wright, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
At this time, IPD will remain anonymous unless a data sharing agreement is made.

REFERENCES:
- [Derived] Bradley SS, de Holanda LJ, Chau T, Wright FV. Physiotherapy-assisted overground exoskeleton use: mixed methods feasibility study protocol quantifying the user experience, as well as functional, neural, and muscular outcomes in children with mobility impairments. Front Neurosci. 2024 Jul 31;18:1398459. doi: 10.3389/fnins.2024.1398459. eCollection 2024. PMID 39145294